CLINICAL TRIAL: NCT02920762
Title: Evaluation of Changes in Prescribing Behavior of ER/LA Opioid Prescribers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ER/LA Opioid REMS Program Companies (RPC) (Industry)
Responsible Party: Sponsor
Other Study IDs: Assessment 7
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Opioid Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (8):
- Buprenorphine
  Interventions: Other: on-interventional study - retrospective database review
- Fentanyl
  Interventions: Other: on-interventional study - retrospective database review
- Hydromorphone HCl
  Interventions: Other: on-interventional study - retrospective database review
- Morphine Sulfate
  Interventions: Other: on-interventional study - retrospective database review
- Morphine Sulfate Beads
  Interventions: Other: on-interventional study - retrospective database review
- Oxycodone HCl
  Interventions: Other: on-interventional study - retrospective database review
- Oxymorphone HCl
  Interventions: Other: on-interventional study - retrospective database review
- Tapentadol
  Interventions: Other: on-interventional study - retrospective database review

INTERVENTIONS:
Other: on-interventional study - retrospective database review

SUMMARY:
A study will be performed to evaluate changes in prescribing behavior of prescribers of ER/LA opioids

DETAILED DESCRIPTION:
A study will be performed to evaluate changes in prescribing behavior of prescribers.

1. For products that are indicated for use in opioid-tolerant patients only (i.e., fentanyl transdermal patches, extended-release hydromorphone pills and extended-release morphine pills >90mg), describe trends in the proportion of prescriptions for these products to opioid-non-tolerant patients in the year preceding the availability of REMS-compliant CE courses and compare the proportion of prescriptions to opioid non-tolerant patients pre- versus post-REMS CE course availability
2. For products whose labels indicate that higher dosage strengths should only be used in opioid-tolerant patients, describe trends in the proportion of prescriptions prescribed to opioid non-tolerant patients with a high starting dosage strength; compare the proportion of prescriptions for such products that are prescribed to opioid non-tolerant patients with a high starting dosage strength pre- versus post-REMS CE course availability
3. Describe trends in the proportion of prescriptions for ER/LA opioids prescribed to patients that have early refills of prescriptions and compare this proportion pre- versus post-REMS CE course availability.
4. Compare the concomitant use of benzodiazepines with ER/LA opioids before and after REMS implementation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects filling a prescription for a product of interest during the specified time period will be included.

Exclusion Criteria:

* None

Max Age: 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects filling a prescription for a product of interest indicated for opioid-tolerant patients, filling prescriptions early and determining concomitant use of products as gathered from the IMS National prescription Audit™ and IMS Health, LifeLink™
Sampling Method: Non-Probability Sample
Enrollment: 5575834 (Estimated)
Dates: Primary Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Monthly volume of opioid-tolerant patients prescribed products indicated for use only in opioid-tolerant patients | Monthly over 54 months
Monthly volume of opioid non-tolerant patients prescribed products indicated for use only in opioid-tolerant patients | Monthly over 54 months
Monthly volume of high-starting dose prescriptions in opioid-tolerant patients | Monthly over 54 months
Monthly volume of high starting dose prescriptions in non-opioid tolerant patients | Monthly over 54 months
Proportion of opioid non-tolerant patients that have high-starting dose prescriptions | Monthly over 54 months
Volume of early refills by monthly patient cohort | Monthly over 54 months
Volume of normal refills (non-early refills) by monthly patient cohort | Monthly over 54 months
Proportion of patients receiving early refills | Monthly over 54 months
Early refill rate by monthly patient cohort | Monthly over 54 months
Monthly volume of patients who are using a REMS product and a Benzodiazepine concomitantly | Monthly over 54 months